CLINICAL TRIAL: NCT00695461
Title: L Plantarum 299v to Patients Undergoing Colon Resection - a Randomized Placebo-Controlled Study
Brief Title: Lactobacillus Plantarum 299v in Colon Surgery
Acronym: Lp 299v
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Skane University Hospital (Other)
Responsible Party: Peter Mangell, MD, Dept of Surgery, Malmö University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: PRO NAT 004
Record Dates: First submitted 2008-06-09; First posted 2008-06-11 (Estimated); Last update posted 2008-06-11 (Estimated); Status verified 2008-06

CONDITIONS: Bacterial Translocation; Inflammation; Cell Proliferation
Keywords: Colorectal surgery; Probiotics; Lactobacillus; Bacterial translocation; Postoperative complications; Inflammatory reaction
MeSH Terms: conditions — Inflammation; Hyperplasia; Postoperative Complications

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Receives Lactobacillus plantarum 299v in an oatmeal drink, at a concentration of 10(9) colony-forming-units/ml, 100 ml per day, starting one week before surgery, finishing 5 days after surgery.
  Interventions: Dietary Supplement: Lactobacillus plantarum 299v in oatmeal drink
- 2 (Placebo Comparator): Receives oatmeal drink, 100 ml per day, starting one week before surgery, finishing 5 days after surgery.
  Interventions: Dietary Supplement: Oatmeal drink

INTERVENTIONS:
Dietary Supplement: Lactobacillus plantarum 299v in oatmeal drink — Bacteria in a concentration of 10(9) CFU/ml
  Arms: 1
Dietary Supplement: Oatmeal drink — Oatmeal drink as in arm 1 but without bacteria added.
  Arms: 2

SUMMARY:
Intestinal pathogenes are often involved in postoperative complications after colon surgery. Probiotic bacteria, i e live bacteria which have beneficial effects on the host when ingested, have been shown to reduce bacterial translocation in animal studies. However, in humans studies results have varied. The purpose with this study was to find whether high doses of Lactobacillus plantarum 299v affects the potentially pathogenic microflora of the gut, bacterial translocation and cell proliferation in patients undergoing planned colon surgery.

ELIGIBILITY:
Inclusion Criteria:

* planned resection of colon for malignant or benign disease
* all ages

Exclusion Criteria:

* unable to understand instructions and perform preoperative intake of study preparation
* rectal surgery
* present or past history of endocarditis
* congenital or acquired valvular heart disease

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2001-01; Primary Completion 2004-06 (Actual); Study Completion 2006-08 (Actual)

PRIMARY OUTCOMES:
Change in intestinal bacterial microflora | Before inclusion, after treatment, during surgery, postoperative day 6, 6 weeks, 6 months

SECONDARY OUTCOMES:
Bacterial translocation | During surgery
Inflammatory response (cytokines) | Preoperative, during operation, 3, 24 an 48 hours postoperastive
Cell proliferation | During surgery
Postoperative complications | One week after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Peter Mangell, MD, Principal Investigator — Dept of Surgery, Malmö University Hospital, Malmö, Sweden
Locations (1):
- Dept of Surgery, Malmö University Hospital, Malmo, Sweden